CLINICAL TRIAL: NCT06848361
Title: Empowering Adults With Diabetes: Achieving Self-management Success Through Data-Driven Behavior Change, Pilot Randomized Control Trial
Brief Title: Helping Adults With Type 2 Diabetes Use Their Health Data for Healthy Diabetes Self-Management
Acronym: MPowerHub
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ann-Marie Rosland (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); The Pittsburgh Foundation (Other)
Responsible Party: Sponsor-Investigator, Ann-Marie Rosland, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY23080053; 1R01DK136788-01A1 (NIH)
Record Dates: First submitted 2025-02-21; First posted 2025-02-27 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Type 2 Diabetes Mellitus; Adult; Glucose Monitoring; Mobile Application; Diabetes Self-Management; Activity Tracker; Continuous Glucose Monitoring; Empowerment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Empowerment | interventions — Fitness Trackers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- MPowerHub (Experimental): Participants will:
  1. Meet with a Diabetes Care and Education Specialist for an initial diabetes self-management education session that will include individualized assessment, education, and coaching on how to set personal diabetes self-management behavior goals and action plans, and follow-up education as needed.
  2. Be trained on how to use assigned study devices (MPowerHub, continuous glucose monitor (CGM), and activity tracker).
  3. Be asked to use assigned study devices (MPowerHub, CGM, and activity tracker) for 4 months.
  Interventions: Device: MPowerHub; Device: Continuous Glucose Monitor (CGM); Device: Activity Monitor
- Continuous Glucose Monitor (CGM) Only (Active Comparator): Participants will:
  1. Meet with a Diabetes Care and Education Specialist for an initial diabetes self-management education session that will include individualized assessment, education, and coaching on how to set personal diabetes self-management behavior goals and action plans, and follow-up education as needed.
  2. Be trained on how to use assigned study device (CGM).
  3. Be asked to use assigned study device (CGM) for 4 months.
  Interventions: Device: Continuous Glucose Monitor (CGM)
- Activity Monitor Only (Active Comparator): Participants will:
  1. Meet with a Diabetes Care and Education Specialist for an initial diabetes self-management education session that will include individualized assessment, education, and coaching on how to set personal diabetes self-management behavior goals and action plans, and follow-up education as needed.
  2. Be trained on how to use assigned study device (activity tracker).
  3. Be asked to use assigned study device (activity tracker) for 4 months.
  Interventions: Device: Activity Monitor

INTERVENTIONS:
Device: MPowerHub — The MPowerHub app allows participants to visualize combined trends from a continuous glucose monitor (CGM) and activity monitor as well as daily self-reports in a display that the participant can customize to overlay the behavioral data they would like to compare to intraday and daily glucose data. Summary data will be displayed over time to allow users to identify potential associations between activity, sleep, stress, diet, and medication adherence and time-in-range and blood glucose variability. Participants receive daily prompts to complete five brief questions about daily health behaviors and two weekly goals/action plans and reflections based on motivational interviewing principles.
  Arms: MPowerHub
Device: Continuous Glucose Monitor (CGM) — A CGM is a wearable device that collects frequent data on glucose levels. It includes an integrated sensor that is inserted under the skin and is connected to a small transmitter that automatically sends information to a smart device, allowing the user to track changes in glucose levels.
  Arms: Continuous Glucose Monitor (CGM) Only; MPowerHub
Device: Activity Monitor — A wearable activity monitor will be used to track activity (e.g., steps) and sleep levels. Data can be viewed on the activity monitor or a smart device.
  Arms: Activity Monitor Only; MPowerHub

SUMMARY:
Day-to-day self-management by adults with type 2 diabetes, including glucose monitoring, taking medications, and healthy habits, is essential to avoid diabetes complications, yet, despite the rapidly expanding availability of wearable glucose and activity monitors, successful self-management remains challenging for many. This research aims to develop and test an approach to help adults use their personal diabetes information from wearable devices to achieve and sustain health diabetes self-management, which will reduce diabetes complications, and improve health and quality of life for people with type 2 diabetes.

DETAILED DESCRIPTION:
MPowerHub trial protocol feasibility will be assessed by randomizing 80 adults with type 2 diabetes and glycemic levels above clinical goals to MPowerHub (MPowerHub platform + continuous glucose monitoring & activity monitoring), continuous glucose monitor alone, or activity monitor alone for four months. Mixed quantitative and qualitative assessments will examine recruitment, engagement, and retention metrics and feedback. Finally, changes in self-management behaviors (measured using semi-structured interview) and clinic glycemic levels (obtained from participants' electronic health record or finger-stick by study research staff) from pre- to post-monitoring will be compared between arms.

ELIGIBILITY:
Inclusion Criteria:

* Received outpatient care in the participating health system in the last 12 months
* Has a diagnosis of type 2 diabetes mellitus (ICD10 codes E08.xx, E09.xx, E11.xx, E13.xx,O24.1x , O24.3x, O24.8x, O24.9x)
* Last Hemoglobin A1c (HbA1c) value obtained in the last 6 months was ≥7.5%
* Currently prescribed at least one non-insulin diabetes medication
* Able to provide informed consent
* Able to interact with a simple smartphone application
* Owns or has access to a smartphone that is able to access an internet website
* Did not participate a prior study related to this protocol

Exclusion Criteria:

* Originally was diagnosed with type 2 diabetes before the age of 21 years
* Has a diagnosis of type 1 diabetes mellitus
* Has a diagnosis of gestational diabetes without any other diabetes diagnoses
* Is currently prescribed insulin
* Currently is using a CGM device
* Has a diagnosis (active or prior) of schizophrenia or other psychotic/delusional disorder
* Has a life-limiting severe illness (e.g., chronic obstructive pulmonary disease requiring oxygen)
* Is pregnant or planning to become pregnant within the next 6 months
* Has other concerns that may interfere significantly with their ability to participate in the intervention (ongoing health issues, personal events, etc.)
* Currently is enrolled in another diabetes management intervention study

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percent of eligible individuals who enroll in the study | Pre-baseline
  Percent of individuals contacted and found eligible who enroll in the study. The goal benchmark is >/=60%.
Percent of days wearable device data is collected | From 0 to 4 months
  Percent of days adequate wearable device data is collected during the 4-month intervention. The goal benchmark is >/=75%.
Percent participants retained in study to the 4-month outcome assessment | From 0 to 4 months
  Percent of participants retained in the study through the 4-month outcome assessment. The goal benchmark is >/=85%.

SECONDARY OUTCOMES:
Percent of individuals contacted who enroll in the study | Pre-baseline
  Percent among all individuals approached/contacted who enroll in the study. The goal benchmark is >/=20%.
Percent of days self-report data is collected | From 0 to 4 months
  Percent of days self-report data is collected from participants in MPowerHub study arm. The goal benchmark is >/=75%.
Percent of weeks participant responds to goal-setting prompts | From 0 to 4 months
  Percent of weeks participants in MPowerHub study arm respond to goal-setting prompts. The goal benchmark is >/=65%.
Participant satisfaction with intervention | 4 months
  Study specific Likert-scaled survey item will be used to assess overall intervention satisfaction by participants. Response options range from 1=highly unsatisfied to 5=highly satisfied. Satisfaction will be defined as a rating of 4=satisfied or 5=highly satisfied. The goal benchmark is >/=80% satisfaction for the MPowerHub arm. The results for MPowerHub arm will also be compared to the two other arms.
Change in hemoglobin A1c | Baseline vs 4-6 Months
  Hemoglobin A1c (HbA1c) data will be obtained from participant's electronic health record. The most recent HbA1c value recorded within 0-6 months prior to enrollment will be used for the baseline measure, and the most recent value recorded at 4-6 months post-enrollment will be used for the outcome measure. If no results from routine HbA1c have been recorded during the relevant time period, the outcome HbA1c data will be collected with a National Glycohemoglobin Standardization Program-certified point of care instrument.
Change in diabetes medication regimen | From baseline to 4-6 months
  Prescribed diabetes medications will be obtained from the participant's electronic health record. A change in diabetes medication regimen assessed by calculating the change in diabetes medication class, e.g., adding or subtracting a class or classes. The range could be negative to positive (e.g., -2, -1, 0, +1, +2) depending on if and how many classes changes occurred.
Started on insulin | From baseline to 4-6 months
  Prescribed insulin during the course of the intervention will be obtained from the participant's electronic health record and documented as yes/no.
Change in medication adherence | Baseline vs. 4 Months
  Medication adherence will be assessed using the self-report Domains of Subjective Extent of Nonadherence (DOSE-Nonadherence) scale, which is comprised of 3 items assessing the extent to which participants missed, skipped, or did not take their medication as prescribed during the past 7 days. Possible scores range from 1=none of the time to 5=every time with a lower score indicating a greater degree of adherence. Items are summed and scores are averaged. The higher the score, the greater the nonadherence.
Change in healthy eating | Baseline vs 4 Months
  Healthy eating will be assessed using the "overall health eating" Summary of Diabetes Self-Care Activities (SDSCA) scale. Participants will be asked how many of the last 7 days have they followed a healthy eating plan (0=no days and 7=all the days). The higher the score, the healthier the eating plan.
Change in fruit and vegetable intake per day | Baseline vs 4 months
  Change in fruit and vegetable intake will be assessed using the 6-item Behavioral Risk Factor Surveillance System (BRFSS) 2017 Fruit and Vegetable Module. Change in daily frequency of fruit and vegetable intake will be calculated using the BRFSS scoring algorithm.
Change in physical activity | Baseline vs 4 Months
  Change in physical activity will be assessed using the International Activity Questionnaire - Short Form (IPAQ-SF). The IPAQ-SF asks respondents to report their frequency and duration of walking, moderate-intensity activity, and vigorous-intensity activity in minutes or hours per day. Our study will score results within each domain separately. Responses will be converted into metabolic equivalent of task (MET) minutes; the higher the MET minutes, the higher the degree of physical activity.
Change in goal setting | Baseline vs 4 months
  Change in goal setting will be assessed using the Patient Assessment of Chronic Illness Care (PACIC) survey. The PACIC includes three questions about thoughts and actions around setting diabetes goals with 5-point Likert scales (almost never to almost always). Scores will be summed from 3 (all almost never) to 15 (all almost always) and averaged with higher scores reflecting better goal setting.
Change in intrinsic motivation | Baseline vs 4 months
  Change in intrinsic motivation will be assessed using the Treatment Self-Regulation Questionnaire (TSRQ) Concerning Diabetes Scale A. The scale includes 3 questions related to autonomous regulation questions measured through a 7-point Likert scale, where 1 is "not at all true", 4 is "somewhat true", and 7 is "very true". Scores will be summed and divided by the total number of items. The higher the score, the higher the level of autonomous regulation.
Change in extrinsic motivation | Baseline vs 4 months
  Change in extrinsic motivation will be assessed using the Treatment Self-Regulation Questionnaire (TSRQ) Concerning Diabetes Scale A. The scale includes 5 questions related to controlled regulation questions measured through a 7-point Likert scale, where 1 is "not at all true", 4 is "somewhat true", and 7 is "very true". Scores will be summed and divided by the total number of items. The higher the score, the higher the level of controlled regulation.
Change in empowerment | Baseline vs 4 months
  Change in empowerment will be assessed using the Diabetes Empowerment Scale-Short Form (DES-SF). Participants will be asked to respond to 8 questions measured through a 5-point Likert scale (strongly disagree to strongly agree). Scores will be summed and divided by the total number of items. The higher the score indicates a higher level of empowerment.
Change in diabetes distress - overall | Baseline vs 4 months
  Change in overall diabetes distress will be assessed using the Diabetes Distress Scale - 17 (DDS17), which yields a total diabetes distress score. To score, participant's responses to the appropriate items are summed and divided by the number of items in the scale (possible range 1-6). The higher the score indicates a higher level of distress.
Change in diabetes distress - emotional burden | Baseline vs 4 months
  Change in emotional burden will be assessed using the Diabetes Distress Scale - 17 (DDS17), which yields a subscale score addressing emotional burden. To score, participant's responses to the appropriate items are summed and divided by the number of items in the emotional burden subscale, possible range 1-6). The higher the score indicates a higher level of distress.
Change in diabetes distress - regimen distress | Baseline vs 4 months
  Change in regimen distress will be assessed using the Diabetes Distress Scale - 17 (DDS17), which yields a subscale score addressing regimen distress. To score, participant's responses to the appropriate items are summed and divided by the number of items in the regimen distress subscale, possible range 1-6). The higher the score indicates a higher level of distress.
Participant rating of intervention usability | 4 months
  Intervention usability will be assessed using the System Usability Scale. Participants will be asked to respond to 10 questions measured through a 5-point Likert scale (strongly disagree to strongly agree). To score, values are converted to 0 to 4 by subtracting one from odd item responses and subtracting 5 from even-numbered items. Converted responses are summed and the total is multiplied by 2.5; the converted range of possible values is from 0 to 100 (with 100 being the most positive response).
Participant perceptions of the benefit of continuous glucose monitoring systems | 4 months
  Perceptions about the benefits of continuous glucose monitoring (CGM) systems will be assessed using the Perceived Benefits of CGM (BenCGM) scale. Participants in the MPowerHub and CGM study arms will be asked 8 questions measured with a 5-point Likert scale (strongly disagree to strongly agree). Item scores are summed and range from 8 (all strongly disagree) to 40 (all strongly agree).
Participant perceptions of the barriers of continuous glucose monitoring systems | 4 months
  Perceptions about the barriers of continuous glucose monitoring (CGM) systems will be assessed using the Perceived Barriers of CGM (BurCGM) scale. Participants in the MPowerHub and CGM study arms will be asked 8 questions measured with a 5-point Likert scale (strongly disagree to strongly agree). Item scores are summed and range from 8 (all strongly disagree) to 40 (all strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Marie Rosland, MD, MS, Principal Investigator — University of Pittsburgh; Carissa Low, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data derived from the trial will be eligible to be shared. Data sets will include only "limited access data" (i.e., no records with personal identifiers). Data sets will be de-identified prior to distribution, and wearable sensor data will be aggregated at a level that is determined to preserve individual confidentiality. Data sharing will follow the NIDDK Policy for Data Sharing (https://niddk.nih.gov/research-funding/research-resources/data-management-sharing).
Supporting Information: Study Protocol, ICF
Time Frame: Data underlying publication will be made available on the study publication date. Data not used in publications will be prepared for sharing by the completion of the award and will remain available for at least five years.
Access Criteria: Data requests must be submitted in writing using a structured data request form. All data requests will be reviewed by the Multiple PIs (MPIs) and subject to the join approval of the MPIs and co-investigators prior to sharing. Requesters will be required to sign a data use agreement prior to receiving access to the data. The requesting institution's IRB or equivalent body must approve the requested use. All data sharing will follow institutional policies and local IRB rules, as well as local, state, and Federal laws and regulations including the HIPAA Privacy Rule.